CLINICAL TRIAL: NCT01283334
Title: A Phase I/IIB Study of Combination Weekly Carboplatin, Cetuximab and Dose Escalation of RAD001 in Recurrent Metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: A Study of Carboplatin, Cetuximab and RAD001 in Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Nabil F. Saba, Physician, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00040298; WCI1761-09 (Other: Other)
Record Dates: First submitted 2011-01-24; First posted 2011-01-25 (Estimated); Results first posted 2014-12-04 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-11

CONDITIONS: Head and Neck Neoplasms; Cancer of the Head and Neck
Keywords: Head and Neck Cancer; Recurrent Metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN)
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Carboplatin; Cetuximab; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Treatment arm with carboplatin, cetuximab and RAD001
  Interventions: Drug: Carboplatin; Drug: Cetuximab; Drug: RAD001

INTERVENTIONS:
Drug: Carboplatin — Will be given as a 30 minutes intravenous (IV) infusion on days 1, 8, and 15 of each 28 day cycle. The starting dose of carboplatin will be area under the plasma-concentration time curve (AUC) = 2 mg/ml.min. Appropriate dose reductions will be done for toxicity for subsequent cycles.
  Other Names: Paraplatin
Drug: Cetuximab — Will be given on days 1, 8, 15 and 22 of each 29 day cycle. On week 1, a loading dose of 400 mg/m² will be given. From week 2 onwards, the dose of cetuximab will be 250 mg/m².
  Other Names: Erbitux
Drug: RAD001 — For phase I, dose escalation will be 2.5 mg, 5 mg, 7.5 mg or 10 mg given orally on a daily basis.
  Other Names: Everolimus; Certican

SUMMARY:
The purpose of this study is to test the drug RAD001 in combination with other chemotherapy drugs, Carboplatin and Cetuximab. Because RAD001 has not been used in this combination before, it is not clear which dose will be best when used in combination.

The investigators will test the safety of RAD001 in combination with Carboplatin and Cetuximab and see what effects (good and/or bad) it has on your cancer, and find the highest dose of RAD001 that can be given without causing bad side effects. The doses of Carboplatin and Cetuximab will not be varied as both these drugs are considered to be part of the current standard of care for patients with your condition.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have at least one measurable site of disease according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria that has not been previously irradiated. If the patient has had previous radiation to the marker lesion(s), there must be evidence of progression since the radiation.
* Histologically or cytologically proven squamous cell carcinoma of the head and neck (SCCHN).
* Patients with recurrent, refractory or metastatic squamous cell carcinoma of oral cavity, oropharynx and larynx, hypopharynx or paranasal sinus, and unknown primary SCCHN who failed to respond to, or relapsed from prior chemoradiotherapy for definitive treatment of disease.
* Evaluable locoregional and/or metastatic disease according to RECIST criteria (see Section 6) that is not appropriate for treatment by primary surgical resection or radiotherapy.
* Patients may not have had prior chemotherapy for recurrent or metastatic disease.
* Patients must not be candidates for curative therapy.
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Life expectancy of ≥ 4 months.
* Adequate bone marrow, liver and renal function as assessed by the following:

  * Hemoglobin ≥ 9.0/dl
  * Absolute-neutrophil count (ANC ) ≥ 1500/mm3
  * Platelet count ≥ 100,000/mm3
  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN (≤ 5 x ULN for patients with liver involvement)
  * International normalized ratio (INR) ≤ 1.5 or a prothrombin time (PT) and partial thromboplastin time (PTT) within normal limits (Anticoagulation is allowed if target INR ≤ 1.5 on a stable dose of warfarin or on a stable dose of low molecular weight (LMW) heparin for > 2 weeks at time of randomization)
  * Creatinine ≤ 1.5 x ULN
* Fasting serum cholesterol ≤ 300 mg/dL OR ≤ 7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
* Women of childbearing potential must have a negative pregnancy test within 7 days prior to first receiving investigational product. Sexually active women of childbearing potential (WOCBP) must use an effective method of birth control during the course of the study, in a manner such that risk of failure is minimized. Prior to study enrollment, WOCBP must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. In addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential and should practice an effective method of birth control. All WOCBP should be instructed to contact the Investigator immediately if they suspect they might be pregnant (e.g., missed or late menstrual period) at any time during study participation.
* Signed informed consent prior to beginning protocol specific procedures. Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care. Patients or their legal representatives must be able to read, understand and provide informed consent to participate in the trial.

Exclusion Criteria:

* History of prior malignancy within the past 5 years except for curatively treated basal cell carcinoma and squamous cell carcinoma of the skin, cervical intraepithelial neoplasia (CIN) or localized prostate cancer with a current prostate-specific antigen (PSA) < 1.0 mg/dL on 2 successive evaluations at least 3 months apart, with the most recent evaluation within 4 weeks of study entry.
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases. Patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude brain metastasis.
* Patients currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks of the start of study drug (including chemotherapy, radiation therapy, antibody based therapy, etc.).
* Prior treatment with any investigational drug within the preceding 4 weeks.
* Any unresolved toxicity (except alopecia) greater than NCI-Common Toxicity Criteria for Adverse Effects (CTCAE) v3.0 grade 2 from prior systemic anticancer therapy.
* Patients who have received prior treatment with a mammalian target of rapamycin (mTOR) inhibitor (sirolimus, temsirolimus, everolimus).
* Patients with a known hypersensitivity to RAD001 (everolimus) or other rapamycins (sirolimus, temsirolimus) or to its excipients, or to cetuximab.
* Prior therapy with Cetuximab will be allowed provided it was part of definitive therapy and not part of treatment for recurrent or metastatic disease.
* Prior severe infusion reaction to a monoclonal antibody.
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent. Topical or inhaled corticosteroids are allowed.
* Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period.
* Patients, who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or patients that may require major surgery during the course of the study.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

  * Symptomatic congestive heart failure of New York heart Association Class III or IV
  * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
  * Severely impaired lung function as defined as spirometry and diffusing capacity of lung for carbon monoxide (DLCO) that is 50% of the normal predicted value and/or 02 saturation that is 88% or less at rest on room air
  * Uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN
  * Active (acute or chronic) or uncontrolled severe infections
  * Liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis
* Abnormal liver function tests (LFTs) as follows: total bilirubin (TB) > 1.5x ULN, alanine aminotransferase (ALT) > 1.25x ULN, and/or alkaline phosphatase > 2.5 x ULN (except when LFTs attributed to metastatic SCCHN, in which case, TB, ALT and alkaline phosphatase must be ≤ NCI-CTCAE, v3.0 grade 1).
* Absolute neutrophil count < 1000/mm3 or platelets < 100,000/mm3.
* A known history of HIV seropositivity.
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection).
* Patients with an active, bleeding diathesis.
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. If barrier contraceptives are being used, these must be continued throughout the trial by both sexes. Hormonal contraceptives are not acceptable as a sole method of contraception. (WOCBP must have a negative urine or serum pregnancy test within 7 days prior to administration of RAD001).
* History of noncompliance to medical regimens.
* Patients unwilling to or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2013-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nabil F. Saba, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States

REFERENCES:
- [Result] Saba NF, Hurwitz SJ, Magliocca K, Kim S, Owonikoko TK, Harvey D, Ramalingam SS, Chen Z, Rogerio J, Mendel J, Kono SA, Lewis C, Chen AY, Higgins K, El-Deiry M, Wadsworth T, Beitler JJ, Shin DM, Sun SY, Khuri FR. Phase 1 and pharmacokinetic study of everolimus in combination with cetuximab and carboplatin for recurrent/metastatic squamous cell carcinoma of the head and neck. Cancer. 2014 Dec 15;120(24):3940-51. doi: 10.1002/cncr.28965. Epub 2014 Aug 7. PMID 25103371

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After institutional review board approval, the study enrolled 20 patients with recurrent or metastatic squamous cell carcinoma of the head and neck (RMSCCHN).
Groups:
- Carboplatin, Cetuximab and Everolimus: Carboplatin, cetuximab and RAD001 (everolimus)
  Carboplatin, cetuximab and RAD001: For phase I, dose escalation will be 2.5mg, 5mg, 7.5mg or 10mg given orally on a daily basis
Period: Overall Study
Arm/Group | Carboplatin, Cetuximab and Everolimus
Started | 20
Completed | 13
Not Completed | 7
Not completed — Withdrawal by Subject | 1
Not completed — Inability to Swallow Everolimus Pills | 1
Not completed — Adverse Event | 4
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Carboplatin, Cetuximab and Everolimus
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: To Measure the Safety and Clinical Effectiveness of the Combination of Carboplatin, Cetuximab and RAD001 in Patients With Advanced (Recurrent or Metastatic) Head and Neck Cancer
Description: This phase 1 clinical trial used a standard 3 + 3 design. Four dose levels of everolimus were planned to be evaluated, and the standard 3 + 3 design with dose de-escalation was used in the trial. Namely, 3 patients were assigned to starting dose level 1. If no dose-limiting toxicity (DLT) was observed, the trial proceeded to the next dose level, and another cohort of 3 patients was enrolled. If at least 2 of the 3 patients experienced at least 1 DLT, then the dose level decreased; otherwise, if only 1 patient experienced DLT, then 3 more patients were enrolled at the same dose level. If none of the 3 additional patients experienced DLT, the dose was escalated; otherwise, the dose level decreased. Dose reduction continued until a dose level was reached at which 6 patients had been treated and at most 1 DLT was observed.
Time Frame: Within the first 21 days of therapy
Measure: Number; unit: participants
Groups:
- Everolimus Dose Level 1 DLT: Carboplatin, cetuximab and RAD001 (everolimus) at Dose Level 1 (2.5 mg/day)
- Everolimus Dose Level -1 DLT: Carboplatin, cetuximab and RAD001 (everolimus) at Dose Level -1 (2.5 mg every other day)
Arm/Group | Everolimus Dose Level 1 DLT | Everolimus Dose Level -1 DLT
Number analyzed (Participants) | 6 | 6
participants | 2 | 1

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Objective tumor responses were assessed every 2 cycles of chemotherapy with computed tomography or positron emission tomography/ computed tomography scans in accordance with Response Evaluation Criteria In Solid Tumors (RECIST) criteria.
Time Frame: The time of PFS was calculated as the time from study enrollment to the disease progression date, death date, or last contact, whichever came first, up to 25 months
Measure: Median (Full Range); unit: months
Arm/Group | Carboplatin, Cetuximab and Everolimus
Number analyzed (Participants) | 13
months | 8.15 [1 to 37]

ADVERSE EVENTS:
Time Frame: Up to 25 months
Arm/Group | Carboplatin, Cetuximab and Everolimus
Serious Adverse Events (participants affected / at risk) | 2/20
Other Adverse Events (participants affected / at risk) | 7/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carboplatin, Cetuximab and Everolimus (N=20)
Nausea and vomiting (Gastrointestinal disorders) | 1 — Patient admitted to emergency department (ED)
Hemoptysis and death (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carboplatin, Cetuximab and Everolimus (N=20)
Neutropenia (Blood and lymphatic system disorders) | 7
Hyperglycemia (Metabolism and nutrition disorders) | 5
Anaphylaxis (Immune system disorders) | 4
Hypokalemia (Blood and lymphatic system disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 4
Hypophosphatemia (Blood and lymphatic system disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3
Fatigue (General disorders) | 2
Hyponatremia (Blood and lymphatic system disorders) | 2
Anemia (Blood and lymphatic system disorders) | 1
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Sepsis (Infections and infestations) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Mucositis (Skin and subcutaneous tissue disorders) | 3
Hypophosphatemia (Blood and lymphatic system disorders) | 6

LIMITATIONS AND CAVEATS:
Limitations of this analysis include the small sample size in this phase 1b study, a patient population with mixed primary sites of disease, and variable doses of everolimus.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes